CLINICAL TRIAL: NCT00916409
Title: A Prospective, Multi-center Trial of NovoTTF-100A Together With Temozolomide Compared to Temozolomide Alone in Patients With Newly Diagnosed GBM.
Brief Title: Effect of NovoTTF-100A Together With Temozolomide in Newly Diagnosed Glioblastoma Multiforme (GBM)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF-14
Record Dates: First submitted 2009-06-05; First posted 2009-06-09 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma Multiforme; Glioblastoma; GBM; Brain tumor; Treatment; Minimal toxicity; Newly Diagnosed; TTFields; Tumor Treating Fields; NovoCure
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NovoTTF-100A device in combination with Temozolomide (Experimental): patients will be treated continuously with the NovoTTF-100A device, in addition to Temozolomide. NovoTTF-100A treatment will consist of wearing four electrically insulated electrode arrays on the head. The treatment enables the patient to maintain regular daily routine.
  Interventions: Device: NovoTTF-100A device
- Temozolomide alone, as the best known standard of care (Active Comparator): Patients will be treated with Temozolomide, as the best known standard of care for Glioblastoma Multiforme patients.
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Device: NovoTTF-100A device — patients will be treated continuously with the NovoTTF-100A device, in addition to Temozolomide. NovoTTF-100A treatment will consist of wearing four electrically insulated electrode arrays on the head. The treatment enables the patient to maintain regular daily routine.
  Arms: NovoTTF-100A device in combination with Temozolomide
Drug: Temozolomide — maintenance Temozolomide will be administered according to the approved dosing scheme as follows: Maintenance Phase Cycle 1: Four weeks after completing the Temozolomide + Radiotherapy phase, Temozolomide is administered for an additional 6 cycles of maintenance treatment. Dosage in Cycle 1 (maintenance) is 150 mg/m2 once daily for 5 days followed by 23 days without treatment.
  Cycles 2-6: At the start of Cycle 2, the dose is escalated to 200 mg/m2, if the CTC non-hematologic toxicity for Cycle 1 is Grade ≤2 (except for alopecia, nausea and vomiting), absolute neutrophil count (ANC) is ≥ 1.5 x 109/L, and the platelet count is ≥ 100 x 109/L. The dose remains at 200 mg/m2 per day for the first 5 days of each subsequent cycle except if toxicity occurs. If the dose was not escalated at Cycle 2, escalation should not be done in subsequent cycles.
  Arms: Temozolomide alone, as the best known standard of care

SUMMARY:
The study is a prospective, randomly controlled pivotal trial, designed to test the efficacy and safety of a medical device, the NovoTTF-100A, as an adjuvant to the best standard of care in the treatment of newly diagnosed GBM patients. The device is an experimental, portable, battery operated device for chronic administration of alternating electric fields (termed TTFields or TTF) to the region of the malignant tumor, by means of surface, insulated electrode arrays.

DETAILED DESCRIPTION:
PAST CLINICAL EXPERIENCE:

The effect of the electric fields generated by the NovoTTF-100A device (TTFields, TTF) has been tested in a large prospective, randomized trial, in recurrent GBM. The outcome of subjects treated with the NovoTTF-100A device was compared to those treated with an effective best standard of care chemotherapy (including bevacizumab). NovoTTF-100A subjects had comparable overall survival to subjects receiving the best available chemotherapy in the US today. Similar results showing comparability of NovoTTF-100A to BSC chemotherapy were seen in all secondary endpoints.

Recurrent GBM patients treated with the NovoTTF-100A device in this trial experienced fewer side effects in general, significantly fewer treatment related side effects, and significantly lower gastrointestinal, hematological and infectious adverse events compared to controls. The only device-related adverse events seen were a mild to moderate skin irritation beneath the device electrodes. Finally, quality of life measures were better in NovoTTF-100A subjects as a group when compared to subjects receiving effective best standard of care chemotherapy.

In a small scale pilot trial in newly diagnosed GBM patients, the treatment was well tolerated and suggested that NovoTTF-100A may improve time to disease progression and overall survival of newly diagnosed GBM patients. Although the number of patients in the pilot trial was small, The FDA has determined that the data gathered so far warrant testing of NovoTTF-100A treatment as a possible therapy for patients with newly diagnosed GBM.

DESCRIPTION OF THE TRIAL:

All patients included in this trial are newly diagnosed GBM patients who underwent a biopsy or surgery (with or without Gliadel wafers), followed by radiation therapy in combination with Temozolomide chemotherapy. In addition, all patients must meet all eligibility criteria.

Eligible patients will be randomly assigned to one of two groups:

1. Treatment with the NovoTTF-100A device in combination with Temozolomide chemotherapy.
2. Treatment with Temozolomide alone, as the best known standard of care.

Patients will be randomized at a 2:1 ratio (2 of every three patients who participate in the trial will be treated with the NovoTTF-100A device). Baseline tests will be performed in patients enrolled in both arms, including specific genetic tests done using tumor samples obtained during their initial surgery. If assigned to the NovoTTF-100A in combination with Temozolomide group, the patients will be treated continuously with the device until second progression. They will also receive temozolomide and possibly a second line treatment that can be one of the following: re-operation, local radiotherapy (gamma-knife), a second line of chemotherapy or a combination of the above.

NovoTTF-100A treatment will consist of wearing four electrically insulated electrode arrays on the head. Electrode array placement will require shaving of the scalp before and frequently during the treatment. After an initial short visit to the clinic for training and monitoring, patients will be released to continue treatment at home where they can maintain their regular daily routine.

During the trial, regardless of which treatment group the patient was assigned to, he or she will need to return once every month to the clinic where an examination by a physician and a routine laboratory examinations will be done. These routine visits will continue for as long as the patient's disease is not progressing for the second time under the study treatment. If such occurs, patients will need to return once per month for two more months to the clinic for similar follow up examinations.

During the visits to the clinic patients will be examined physically and neurologically. Additionally, routine blood tests will be performed. A routine MRI of the head will be performed at baseline and every second month thereafter, until second progression. After this follow up plan, patients will be contacted once per month by telephone to answer basic questions about their health status.

SCIENTIFIC BACKGROUND:

Electric fields exert forces on electric charges similar to the way a magnet exerts forces on metallic particles within a magnetic field. These forces cause movement and rotation of electrically charged biological building blocks, much like the alignment of metallic particles seen along the lines of force radiating outwards from a magnet.

Electric fields can also cause muscles to twitch and if strong enough may heat tissues. TTFields are alternating electric fields of low intensity. This means that they change their direction repetitively many times a second. Since they change direction very rapidly (200 thousand times a second), they do not cause muscles to twitch, nor do they have any effects on other electrically activated tissues in the body (brain, nerves and heart). Since the intensities of TTFields in the body are very low, they do not cause heating.

The breakthrough finding made by NovoCure was that finely tuned alternating fields of very low intensity, now termed TTFields (Tumor Treating Fields), cause a significant slowing in the growth of cancer cells. Due to the unique geometric shape of cancer cells when they are multiplying, TTFields cause the building blocks of these cells to move and pile up in such a way that the cells physically explode. In addition, cancer cells also contain miniature building blocks which act as tiny motors in moving essential parts of the cells from place to place. TTFields cause these tiny motors to fall apart since they have a special type of electric charge.

As a result of these two effects, cancer tumor growth is slowed and can even reverse after continuous exposure to TTFields.

Other cells in the body (normal healthy tissues) are affected much less than cancer cells since they multiply at a much slower rate if at all. In addition TTFields can be directed to a certain part of the body, leaving sensitive areas out of their reach.

In conclusion, TTField hold the promise of serving as a brand new cancer treatment with very few side effects and promising affectivity in slowing or reversing this disease.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological evidence of GBM using WHO classification criteria.
2. > 18 years of age.
3. Received maximal debulking surgery and radiotherapy concomitant with Temozolomide (45-70Gy):

   1. Patients may enroll in the study if received Gliadel wafers before entering the trial
   2. Any additional treatments received prior to enrollment will be considered an exclusion.
   3. Minimal dose for concomitant radiotherapy is 45 Gy
4. Karnofsky scale ≥ 70
5. Life expectancy at least 3 months
6. Participants of childbearing age must use effective contraception.
7. All patients must sign written informed consent.
8. Treatment start date at least 4 weeks out from surgery.
9. Treatment start date at least 4 weeks out but not more than 7 weeks from the later of last dose of concomitant Temozolomide or radiotherapy.

Exclusion Criteria:

1. Progressive disease (according to MacDonald Criteria). If pseudoprogression is suspected, additional imaging studies must be performed to rule out true progression.
2. Actively participating in another clinical treatment trial
3. Pregnant
4. Significant co-morbidities at baseline which would prevent maintenance Temozolomide treatment:

   1. Thrombocytopenia (platelet count < 100 x 103/μL)
   2. Neutropenia (absolute neutrophil count < 1.5 x 103/μL)
   3. CTC grade 4 non-hematological Toxicity (except for alopecia, nausea, vomiting)
   4. Significant liver function impairment - AST or ALT > 3 times the upper limit of normal
   5. Total bilirubin > upper limit of normal
   6. Significant renal impairment (serum creatinine > 1.7 mg/dL)
5. Implanted pacemaker, programmable shunts, defibrillator, deep brain stimulator, other implanted electronic devices in the brain, or documented clinically significant arrhythmias.
6. Infra-tentorial tumor
7. Evidence of increased intracranial pressure (midline shift > 5mm, clinically significant papilledema, vomiting and nausea or reduced level of consciousness)
8. History of hypersensitivity reaction to Temozolomide or a history of hypersensitivity to DTIC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2009-06; Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) time | 5 years

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Roger Stupp, MD, Study Director — University Hospital, Zürich; Philip H. Gutin, MD, Study Director — Memorial Sloan Kettering Cancer Center; Eric T. Wong, MD, Study Director — Beth Israel Deaconess Medical Center; Herbert H. Engelhard, MD, PhD, Study Director — University of Illinois at Chicago; Manfred Westphal, Prof. MD, Study Director — Universitätsklinikum Hamburg-Eppendorf
Locations (89):
- United States (41):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Barrow Neurology Clinics, Phoenix, Arizona
  - City of Hope, Duarte, California
  - University of California San Diego Moores Cancer Center (UCSD), La Jolla, California
  - University of Southern California (USC), Los Angeles, California
  - University of Colorado Denver, Aurora, Colorado
  - UF Health Cancer Center at Orlando Health, Orlando, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Emory University, Winship Cancer Institute, Atlanta, Georgia
  - University of Illinois at Chicago (UIC), Chicago, Illinois
  - University of Kentucky, Markey Cancer Center, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Maine Medical Center, Scarborough, Maine
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Washington University School of Medicine, Division of Oncology, St Louis, Missouri
  - New Jersey Neuroscience Center - JFK Medical Center, Edison, New Jersey
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Weill Cornell Medical College, New York, New York
  - Mount Sinai Medical Center, Department of Neurosurgery, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - The Ohio State University Arthur G. James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - Geisinger Health System, Danville, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor, Dallas, Texas
  - Methodist Hospital, Houston, Texas
  - Methodist Neurological Institute, Houston, Texas
  - The University of Texas Health Science Center at Houston (UTHSC), Houston, Texas
  - Scott and White Healthcare, Temple, Texas
  - Memorial Hermann The Woodlands, The Woodlands, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Swedish Neuroscience Institute, Seattle, Washington
  - University of Washington/Seattle Cancer Care Alliance, Seattle, Washington
- Austria (3):
  - University Hospital Graz, Graz
  - Medical University of Vienna, Vienna
  - SMZ-Süd/Kaiser-Franz-Josef-Spital, Vienna
- Canada (8):
  - Tom Baker Cancer Center, Calgary, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Juravinski Cancer Centre, Hamilton, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Notre-Dame Hospital (CHUM), Montreal, Quebec
  - Montreal Neurological Institute, Montreal, Quebec
  - McGill - Gerald Bronfman Centre for Clinical Research in Oncology -, Montreal, Quebec
  - (CHUS) Centre Hospitalier Universitaire de Sherbrooke, Service de Neurochirurgie, Sherbrooke, Quebec
- Na Homolce Hospital, Prague, Czechia
- France (6):
  - CHU Amiens Sud-Salouel, Amiens
  - CHU Angers, Angers
  - Hôpital Saint André Centre Hospitalier Universitaire (CHU) des Hôpitaux de Bordeaux, Bordeaux
  - Hospital of Neurology Pierre Wertheimer, Lyon
  - Group Hospitals Pitie-Salpetriere, Paris
  - Centre Hospitalo-Universitaire de Toulouse Purpan, Toulouse
- Germany (3):
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Medical University Heidelberg, Heidelberg
  - University Hospital of Schleswig-Holstein, Kiel
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Italy (5):
  - Az. Ospedaliero-Universitaria - Ospedali Riuniti, Ancona
  - Ospedale Lecco, Lecco
  - C. Besta Neurological Institute, Milan
  - Foundation Hospital Greater Policlinico, Milan
  - Istituti Fisioterapici Ospitalieri - Istituto Nazionale dei Tumori Regina Elena, Rome
- South Korea (9):
  - Asan Medical Center, Asan
  - Yeungnam University Hospital, Daegu
  - Chungnam National University Hospital (CNUH), Daejeon
  - Samsung Medical Center (SMC), Seoul
  - Seoul National University Bundang Hospital (SNUBH), Seoul
  - Seoul National University Hospital (SNUH), Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital (CMC Seoul), Seoul
  - Yonsei University Severance Hospital (YUHS), Seoul
  - Ajou University Hospital (AUH), Suwon
- Spain (9):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitari de Bellvitge-ICO Duran i Reynals, Barcelona
  - Fundacion Jimenes Diaz, Madrid
  - Hospital 12 de Octubre, Servicio de Oncología Médica, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Clínica Universidad de Navarra, Pamplona
- Karolinska Institute, Stockholm, Sweden
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne
  - UniversitätsSpital Zürich, Zurich

REFERENCES:
- [Background] Kirson ED, Gurvich Z, Schneiderman R, Dekel E, Itzhaki A, Wasserman Y, Schatzberger R, Palti Y. Disruption of cancer cell replication by alternating electric fields. Cancer Res. 2004 May 1;64(9):3288-95. doi: 10.1158/0008-5472.can-04-0083. PMID 15126372
- [Background] Kirson ED, Dbaly V, Tovarys F, Vymazal J, Soustiel JF, Itzhaki A, Mordechovich D, Steinberg-Shapira S, Gurvich Z, Schneiderman R, Wasserman Y, Salzberg M, Ryffel B, Goldsher D, Dekel E, Palti Y. Alternating electric fields arrest cell proliferation in animal tumor models and human brain tumors. Proc Natl Acad Sci U S A. 2007 Jun 12;104(24):10152-7. doi: 10.1073/pnas.0702916104. Epub 2007 Jun 5. PMID 17551011
- [Background] Salzberg M, Kirson E, Palti Y, Rochlitz C. A pilot study with very low-intensity, intermediate-frequency electric fields in patients with locally advanced and/or metastatic solid tumors. Onkologie. 2008 Jul;31(7):362-5. doi: 10.1159/000137713. Epub 2008 Jun 24. PMID 18596382
- [Background] Kirson ED, Giladi M, Gurvich Z, Itzhaki A, Mordechovich D, Schneiderman RS, Wasserman Y, Ryffel B, Goldsher D, Palti Y. Alternating electric fields (TTFields) inhibit metastatic spread of solid tumors to the lungs. Clin Exp Metastasis. 2009;26(7):633-40. doi: 10.1007/s10585-009-9262-y. Epub 2009 Apr 23. PMID 19387848
- [Background] Kirson ED, Schneiderman RS, Dbaly V, Tovarys F, Vymazal J, Itzhaki A, Mordechovich D, Gurvich Z, Shmueli E, Goldsher D, Wasserman Y, Palti Y. Chemotherapeutic treatment efficacy and sensitivity are increased by adjuvant alternating electric fields (TTFields). BMC Med Phys. 2009 Jan 8;9:1. doi: 10.1186/1756-6649-9-1. PMID 19133110
- [Derived] Ram Z, Kim CY, Hottinger AF, Idbaih A, Nicholas G, Zhu JJ. Efficacy and Safety of Tumor Treating Fields (TTFields) in Elderly Patients with Newly Diagnosed Glioblastoma: Subgroup Analysis of the Phase 3 EF-14 Clinical Trial. Front Oncol. 2021 Sep 27;11:671972. doi: 10.3389/fonc.2021.671972. eCollection 2021. PMID 34692470
- [Derived] Kim CY, Paek SH, Nam DH, Chang JH, Hong YK, Kim JH, Kim OL, Kim SH. Tumor treating fields plus temozolomide for newly diagnosed glioblastoma: a sub-group analysis of Korean patients in the EF-14 phase 3 trial. J Neurooncol. 2020 Feb;146(3):399-406. doi: 10.1007/s11060-019-03361-2. Epub 2020 Feb 4. PMID 32020470
- [Derived] Ballo MT, Urman N, Lavy-Shahaf G, Grewal J, Bomzon Z, Toms S. Correlation of Tumor Treating Fields Dosimetry to Survival Outcomes in Newly Diagnosed Glioblastoma: A Large-Scale Numerical Simulation-Based Analysis of Data from the Phase 3 EF-14 Randomized Trial. Int J Radiat Oncol Biol Phys. 2019 Aug 1;104(5):1106-1113. doi: 10.1016/j.ijrobp.2019.04.008. Epub 2019 Apr 23. PMID 31026557
- [Derived] Toms SA, Kim CY, Nicholas G, Ram Z. Increased compliance with tumor treating fields therapy is prognostic for improved survival in the treatment of glioblastoma: a subgroup analysis of the EF-14 phase III trial. J Neurooncol. 2019 Jan;141(2):467-473. doi: 10.1007/s11060-018-03057-z. Epub 2018 Dec 1. PMID 30506499
- [Derived] Taphoorn MJB, Dirven L, Kanner AA, Lavy-Shahaf G, Weinberg U, Taillibert S, Toms SA, Honnorat J, Chen TC, Sroubek J, David C, Idbaih A, Easaw JC, Kim CY, Bruna J, Hottinger AF, Kew Y, Roth P, Desai R, Villano JL, Kirson ED, Ram Z, Stupp R. Influence of Treatment With Tumor-Treating Fields on Health-Related Quality of Life of Patients With Newly Diagnosed Glioblastoma: A Secondary Analysis of a Randomized Clinical Trial. JAMA Oncol. 2018 Apr 1;4(4):495-504. doi: 10.1001/jamaoncol.2017.5082. PMID 29392280
- [Derived] Stupp R, Taillibert S, Kanner A, Read W, Steinberg D, Lhermitte B, Toms S, Idbaih A, Ahluwalia MS, Fink K, Di Meco F, Lieberman F, Zhu JJ, Stragliotto G, Tran D, Brem S, Hottinger A, Kirson ED, Lavy-Shahaf G, Weinberg U, Kim CY, Paek SH, Nicholas G, Bruna J, Hirte H, Weller M, Palti Y, Hegi ME, Ram Z. Effect of Tumor-Treating Fields Plus Maintenance Temozolomide vs Maintenance Temozolomide Alone on Survival in Patients With Glioblastoma: A Randomized Clinical Trial. JAMA. 2017 Dec 19;318(23):2306-2316. doi: 10.1001/jama.2017.18718. PMID 29260225
- [Derived] Kesari S, Ram Z; EF-14 Trial Investigators. Tumor-treating fields plus chemotherapy versus chemotherapy alone for glioblastoma at first recurrence: a post hoc analysis of the EF-14 trial. CNS Oncol. 2017 Jul;6(3):185-193. doi: 10.2217/cns-2016-0049. Epub 2017 Apr 12. PMID 28399638
- [Derived] Meletath SK, Pavlick D, Brennan T, Hamilton R, Chmielecki J, Elvin JA, Palma N, Ross JS, Miller VA, Stephens PJ, Snipes G, Rajaram V, Ali SM, Melguizo-Gavilanes I. Personalized Treatment for a Patient With a BRAF V600E Mutation Using Dabrafenib and a Tumor Treatment Fields Device in a High-Grade Glioma Arising From Ganglioglioma. J Natl Compr Canc Netw. 2016 Nov;14(11):1345-1350. doi: 10.6004/jnccn.2016.0145. PMID 27799506
- [Derived] Stupp R, Taillibert S, Kanner AA, Kesari S, Steinberg DM, Toms SA, Taylor LP, Lieberman F, Silvani A, Fink KL, Barnett GH, Zhu JJ, Henson JW, Engelhard HH, Chen TC, Tran DD, Sroubek J, Tran ND, Hottinger AF, Landolfi J, Desai R, Caroli M, Kew Y, Honnorat J, Idbaih A, Kirson ED, Weinberg U, Palti Y, Hegi ME, Ram Z. Maintenance Therapy With Tumor-Treating Fields Plus Temozolomide vs Temozolomide Alone for Glioblastoma: A Randomized Clinical Trial. JAMA. 2015 Dec 15;314(23):2535-43. doi: 10.1001/jama.2015.16669. PMID 26670971